CLINICAL TRIAL: NCT06251297
Title: Feasibility and Benefits of Reflexology in the Prevention of Neuropathy Induced by Oxaliplatin in Colorectal Cancer
Acronym: FIRENOX
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: RC31/22/0041
Record Dates: First submitted 2024-01-25; First posted 2024-02-09 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Colorectal Cancer
Keywords: oxaliplatin; reflexology
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: All patients will receive a 30-minute reflexology session during each Oxaliplatin infusion.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Reflexology session (Experimental): Patients included in the study and treated with oxaliplatin based regiment will receive 30-min of a standard reflexology session during each infusion for a maximum of 12 sessions over 6 months).
  Interventions: Other: Foot reflexology

INTERVENTIONS:
Other: Foot reflexology — 30 minutes reflexology session

SUMMARY:
The management of colorectal cancer often requires oxaliplatin-based chemotherapy, either as part of curative treatment plans or exclusively in palliative situations. Oxaliplatin therefore plays a key role in the management of colorectal cancer. In addition to its digestive and hematological toxicity, oxaliplatin frequently induces chronic, often limiting, sensitive peripheral neuropathy.

Only early discontinuation of oxaliplatin can limit the risk of clinically limiting neurotoxicity (grade ≥ 3).

In oncology, managing the side-effects of treatment is an essential objective of supportive care, and is open to a variety of complementary medicines, including reflexology. This technique, derived from traditional Chinese medicine, involves stimulating reflex points on the arch of the foot.

DETAILED DESCRIPTION:
This first monocentric, prospective pilot study is designed to evaluate if the intervention is feasible in routine clinical practice for patients initiating bimonthly oxaliplatin chemotherapy for colorectal cancer. It will also provide initial estimates of the parameters needed to measure efficacy and impact on patient quality of life.

Patients will receive a reflexology session with each cycle of chemotherapy, and will be assessed during all the treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Age>18 years treated for colorectal cancer in Digestive Oncology service Rangueil hospital
* Initiation of intravenous oxaliplatin chemotherapy at 85 mg/m² on a bimonthly schedule.
* Ability to understand and answer a self-questionnaire.
* Life expectancy egal or over 12 weeks
* Signed informed consent form

Exclusion Criteria:

* Pre-existing motor and/or sensitive neuropathy.
* Reflexology treatment within the last 6 months.
* Contraindication to reflexology: venous thrombosis, trauma, wound or metastasis of the foot.
* Patient covered by a legal protection scheme.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-04-29 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
number of sessions performed | 6 months
  at least 50% of patients included and realized at least 70% of reflexology sessions over the 6-month treatment.

SECONDARY OUTCOMES:
concordance of peripheral neuropathy evaluation | every month until 6 months
  peripheral neuropathy evaluation between physician's assessment and programming nurse's assessment

CONTACTS AND LOCATIONS:
Overall Officials: Nadim FARES, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- CHU de Toulouse, Toulouse, CHU de Toulouse, France

IPD SHARING:
Plan to Share IPD: No